CLINICAL TRIAL: NCT06243302
Title: Anal Fistulae Internal Opening Closure by OTSC Clip After Video Assisted Tract Fulguration
Acronym: VAAFT-OTSC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, I Ethem Gecim, Prof Dr, Ankara University
Other Study IDs: KRKAP-002
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Anal Fistula
Keywords: VAAFT; OTSC; diathermy Ablation of Fistula Tract
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment Arm: VAAFT followed by OTSC clip inserted to close the inner opening of the anal fistula
  Interventions: Procedure: OTSC Closure After VAAFT

INTERVENTIONS:
Procedure: OTSC Closure After VAAFT — Under general anesthesia,the fistulas will be drained at least for 8 weeks. Then a video camera will be inserted through the external opening to fulgurate the fistula tract under direct vision. Finally the internal fistula opening will be closed water tight by a circular clip. The patients will be followed up for complications as well as short and long term recurrences

SUMMARY:
This study is expected to recruit 20-25 cases treated with video assisted anal fistula treatment. Additionally the internal opening of the fistulae will be closed by an OTSC clip.

DETAILED DESCRIPTION:
Sphincter damage after anal fistulae surgery is the most important cause of incontinence in adults. Surgeons are gradually gradually getting more reluctant for creating any damage to sphincter for this reason. Anteriorly located, high and trans-sphincteric fistulae are at more risk.

Ablating the fistula tract by laser or diathermy has been in use for a long time. Recently a rigid thin camera to visualize all side tracts and branches for ablating them under direct vision has also been in use especially in Europe. Recently, closing the internal opening after ablating the fistula tract was reported to offer higher success rates for healing with less recurrence. The success rate was higher when the opening was closed by a stapler device.

Our aim in this study is to use o novel technique by using OTSC clip for water tight closure of the internal fistula opening after diathermy ablation of the tract under direct vision and compare the healing and recurrence rates with other methods.

ELIGIBILITY:
Inclusion Criteria: Patients with trans-sphincteric and inter-sphincteric perianal fistulae

-

Exclusion Criteria:

* Presence of acute abscess, Inflammatory Bowel Disease, Myeloproliferative disease, established incontinence, Recto-vaginal fistula

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and females with trans-sphincteric perianal fistulas
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2024-02-20 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Fistula healing | January 2024
  No leakage at all

SECONDARY OUTCOMES:
Recurrence | January 2024
  No re-occuring symptoms
perianal abscess/fistula | January 2024
  re-occuring abscess or fistula

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Hospital,Dept of Surgery, Cebeci, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Present it in the ESCP Meeting
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: September 2024
Access Criteria: Primary and secondary outcomes

REFERENCES:
- [Background] Meinero P, Mori L, Gasloli G. Video-assisted anal fistula treatment: a new concept of treating anal fistulas. Dis Colon Rectum. 2014 Mar;57(3):354-9. doi: 10.1097/DCR.0000000000000082. PMID 24509459